CLINICAL TRIAL: NCT02421068
Title: Pharmacokinetic and Pharmacodynamic Modelling of Routinely Used Off Label Drugs in Premature Neonates
Brief Title: Population PK/PD of Off Label Drugs in Premature Neonates
Acronym: DINO
Status: Completed | Type: Observational
Sponsor: Sinno H.P. Simons (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Leiden Amsterdam Centre for Drug Research (LACDR) (Unknown); Dutch Knowledge Centre for Pediatric Pharmacotherapy (NKFK) (Unknown); Centre for Human Drug Research, Netherlands (Other); Radboud University Medical Center (Other)
Responsible Party: Sponsor-Investigator, Sinno H.P. Simons, MD PhD, Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Other Study IDs: NL-47440907814
Record Dates: First submitted 2014-09-25; First posted 2015-04-20 (Estimated); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Premature Birth
Keywords: Paracetamol; Fentanyl; Phenobarbital; Doxapram; Midazolam; Sildenafil; Levetiracetam; Pharmacokinetics; Pharmacology; Fluconazole; Ibuprofen
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Preterm neonates: All neonates that receive at least one of the 9 drugs (phenobarbital, paracetamol, levetiracetam, midazolam, sildenafil, fentanyl, doxapram, ibuprofen, fluconazole) are included in the studied cohort

SUMMARY:
This study will provide information on the pharmacokinetics, safety and effectiveness of off--label drugs used in critically ill premature infants: doxapram, fentanyl, midazolam, paracetamol, phenobarbital, sildenafil, levetiracetam, ibuprofen and fluconazole. PK/PD analysis with NONMEM (non-linear mixed effects modelling) will result in (adapted) dosage guidelines, thus contributing towards an improvement in the quality of care and cost efficiency. Furthermore the development of Dried Blood Spot (DBS) analysis is investigated for these drugs as a minimally invasive method for conventional patient care and to perform pharmacological studies in children. The adapted dosage guidelines will be implemented directly into clinical practice in collaboration with the NKFK. Therefore the study is designed as an observational multicenter study to be able to collect sufficient data for the drugs of interest.

DETAILED DESCRIPTION:
BACKGROUND Approximately 60% of drugs are used off--label in critically ill neonates in the Neonatal Intensive Care Units (NICU). This is even more true for pre--term born neonates in whom pharmacokinetics of these agents may be different due to immature elimination pathways. The lack of sufficient data about efficacy and safety of many of these drugs makes it difficult to have evidence based dosing guidelines for these agents. Therefore the urge for drug research in this population is of great importance. The pharmacokinetic (PK) and pharmacodynamic (PD) characteristics of drugs in premature infants are different from the characteristics found in term neonates, older children and adults. These differences are caused among others by a different body composition, by immaturity of the renal excretion systems, the metabolic pathways in the liver and other organ functions as well as immature drug receptors and transporters. After birth, there is a rapid development of many of these functions, necessitating frequent adaptation of dosage guidelines in the first few weeks of life. Besides age and size, co--morbidity, co--administration of drugs and genetic heterogeneity may further contribute to this extensive inter--individual variability in pharmacokinetics and pharmacodynamics of premature infants. There is a critical lack of evidence--based data of drug dosing in (extremely) preterm neonates.

OBJECTIVE Recently, population PK/PD modeling and simulation studies have enabled the development of evidence--based individualized dosing schemes for children with a limited number of subjects, thus improving drug safety and efficacy. The application of PK/PD modeling in the most critically ill population of premature infants, with the highest variability in the pharmacokinetics of drugs, and the greatest lack of adequate data underscoring optimal dosage, can contribute to the development of rational, individualized and safe dosing regimens.

This study will provide information on the pharmacokinetics, safety and effectiveness of off--label drugs used in critically ill premature infants: doxapram, fentanyl, midazolam, paracetamol, phenobarbital, sildenafil, levetiracetam, ibuprofen and fluconazole (only studied for the PK). PK/PD analysis will result in (adapted) dosage guidelines, thus contributing towards an improvement in the quality of care and cost efficiency. Furthermore the development of Dried Blood Spot (DBS) analysis is investigated for these drugs as a minimally invasive method for conventional patient care and to perform pharmacological studies in children. The adapted dosage guidelines will be implemented directly into clinical practice in collaboration with the NKFK. Therefore the study is designed as an observational multicenter study to be able to collect sufficient data for the drugs of interest.

DESIGN This is a prospective observational multicenter study on the pharmacokinetics and pharmacodynamics of paracetamol, fentanyl, midazolam, phenobarbital, doxapram, levetiracetam, sildenafil, ibuprofen and fluconazole routinely administered to preterm infants according to standard protocols. The treatment regimen is left to the discretion of the treating physician in accordance with current guidelines. During this study a limited number of additional blood samples will be drawn from the participants for pharmacokinetic analysis, never exceeding 3% of the total blood volume during any four--week period or 1% at any single time.

It is standard care in the Netherlands for all premature born infants under 32 weeks to get seen by the paediatrician at the age of two years for a check on growth and development. The visit to the day care clinic of the hospital of their admission on birth, enables us to collect qualitative data on growth and physiological development as well as from psychological and neurodevelopmental standardised tests.The collected data enables us to gain a better description of the subjects in our study and to further determine safety of the studied drugs.

POPULATION All preterm infants born with gestational age < 32 weeks who are admitted to one of the participating NICUs are eligible for inclusion. The participating departments are all level III Neonatal Intensive Care Units. Three are situated in an academic hospital (Rotterdam, Nijmegen and Maastricht) and one in a non--academic hospital (Veldhoven). Patients admitted to the 4 NICUs consist of both inborn and outborn neonates with different gestational ages (24--42 weeks). All admitted patients need intensive or high care treatment. Most patients will be admitted on the first postnatal day, but sometimes are referred at older post natal ages (<14 days) to the NICU.

OUTCOME

Primary study parameters/outcome of the study:

1) Pharmacokinetic endpoints for all 9 drugs are clearance en volume of distribution.

Secondary study parameters/outcome of the study (if applicable):

Pharmacodynamics of paracetamol, fentanyl, midazolam, phenobarbital, doxapram, levetiracetam and sildenafil will be explored in all included preterm neonates. Fluconazole will only be studied for the pharmacokinetics. Drug specific effects of drugs (e.g. pain scores for morphine, blood pressure for dopamine) as well as side effects and short term effects on morbidity and outcome will be analyzed. Additional pharmacodynamic endpoints for the 7 PK/PD study drugs is the drug target concentration for each drug that is related to the desired effect.

The parameters to measure the effect of the drugs:

1. Fentanyl and paracetamol, used as analgetics; clinical endpoint is pain relief, as routinely measured by the validated COMFORTneo scale and the NRS (numeric rating scale) scale.
2. Midazolam, phenobarbital and levetiracetam, used as anticonvulsive drugs; clinical endpoint is control of convulsions, measured by Cerebral Function Monitoring using amplitude--integrated EEG (aEEG).
3. Midazolam and fentanyl, used as a sedative drug during endotracheal intubation; clinical endpoint is the intubation readiness score (IRS) and a qualitative intubation score and sedation score.
4. Midazolam and fentanyl, used as a sedative drug during nursing care is measured by the COMFORTneo scale.
5. Doxapram, used as treatment for neonatal apnea; clinical endpoint is control of neonatal apnea and endotracheal intubation in case of failure. The first endpoint can be measured by modern monitoring technology, in which central post--monitoring data stored after initiation of treatment will reveal the effect of doxapram on the reduction or elimination of apneas.
6. Sildenafil, a treatment for PH (pulmonary hypertension); clinical endpoints are level of ventilatory support, oxygen need (repetitive oxygenation index analyses) and BPD (broncho pulmonary dysplasia) development.
7. Ibuprofen is used to close patent ductus arteriosus (PDA) in different dosages, orally and intravenously in the recruiting sites. Endpoints are measured by cardiac ultrasound: ductus closure (yes/no), ductal diameter and LA/AO ratio

Inter-- and intra--patient variability of the PD and PK parameters of the drugs to be investigated. Parameters with effect on this variability will be identified.

Tertiary outcome:

1. Development of a minimally invasive Dried Blood Spot analysis method to perform future pharmacokinetic studies in neonates. The measured concentration of the drugs in the dried blood spot samples will be compared with the concentration of the blood samples in the vial, which is the current validated standard method. The validity of the DBS method will be the endpoint.
2. Influence of specific polymorphisms involved in the metabolism of the investigated drugs.

ELIGIBILITY:
Inclusion Criteria:

* prescription of one of the seven drug of interest
* parental informed consent

Exclusion Criteria:

- none

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: preterm newborn infants
Sampling Method: Non-Probability Sample
Enrollment: 246 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Clearance, Volume of distribution and covariates for the variability of paracetamol, fentanyl, midazolam, phenobarbital, doxapram, sildenafil, levetiracetam, ibuprofen, and fluconazole in premature born neonates | Participants will be followed for the duration of admission to the NICU, an expected average of 9 weeks. Note that registration and blood sampling only take place when a study drug is being administered
  Clearance, Volume of distribution and variability in premature born neonates will be calculated by population modelling (NONMEM) of the collected data: drug dosages(mg/kg), measured plasmaconcentrations (mg/L) and their metabolites, and patientcharacteristics (body weight, post natal age, gestational age, renal function, gender)

SECONDARY OUTCOMES:
EC50 of midazolam on treatment of convulsions | Participants will be followed for the duration of admission to the NICU, an expected average of 9 weeks. Note that registration and blood sampling only take place when a study drug is being administered
  EC50 describes the relationship between the midazolam concentration and the effect on convulsions at the aEEG, and will be calculated by population modelling (NONMEM)
EC50 of phenobarbital on treatment of convulsions | Participants will be followed for the duration of admission to the NICU, an expected average of 9 weeks. Note that registration and blood sampling only take place when a study drug is being administered
  EC50 describes the relationship between the phenobarbital concentration and the effect on convulsions at the aEEG, and will be calculated by population modelling (NONMEM)
EC50 of levetiracetam on treatment of convulsions | Participants will be followed for the duration of admission to the NICU, an expected average of 9 weeks. Note that registration and blood sampling only take place when a study drug is being administered
  EC50 describes the relationship between the levetiracetam concentration and the effect on convulsions at the aEEG, and will be calculated by population modelling (NONMEM)
EC50 of fentanyl as analgetic | Participants will be followed for the duration of admission to the NICU, an expected average of 9 weeks. Note that registration and blood sampling only take place when a study drug is being administered
  EC50 describes the relationship between the fentanyl concentration and the effect on analgesia measures with the COMFORTneo score, and will be calculated by population modelling (NONMEM)
EC50 of paracetamol as analgetic | Participants will be followed for the duration of admission to the NICU, an expected average of 9 weeks. Note that registration and blood sampling only take place when a study drug is being administered
  EC50 describes the relationship between the paracetamol concentration and the effect on analgesia measures with the COMFORTneo score, and will be calculated by population modelling (NONMEM)
EC50 of fentanyl as sedative drug during endotracheal intubation | Participants will be followed for the duration of admission to the NICU, an expected average of 9 weeks. Note that registration and blood sampling only take place when a study drug is being administered
  EC50 describes the relationship between the paracetamol concentration and the effect on analgesia measures with the COMFORTneo score, and will be calculated by population modelling (NONMEM)clinical endpoint is the intubation readiness score (IRS) and a qualitative intubation score and sedation score.
EC50 of fentanyl as sedative drug during nursing care | Participants will be followed for the duration of admission to the NICU, an expected average of 9 weeks. Note that registration and blood sampling only take place when a study drug is being administered
  level of sedation measured by the COMFORTneo scale during nursing. Outcome measure COMFORTneo 6 - 30
EC50 of midazolam as sedative drug during nursing care | Participants will be followed for the duration of admission to the NICU, an expected average of 9 weeks. Note that registration and blood sampling only take place when a study drug is being administered
  level of sedation measured by the COMFORTneo scale during nursing. Outcome measure COMFORTneo 6 - 30
EC50 of doxapram as treatment for neonatal apnea | Participants will be followed for the duration of admission to the NICU, an expected average of 9 weeks. Note that registration and blood sampling only take place when a study drug is being administered
  control of neonatal apnea (reduction or elimination of apneas) using modern monitoring technology, and endotracheal intubation in case of failure. Outcome measure: Yes or No
EC50 of sildenafil as treatment for PH | Participants will be followed for the duration of admission to the NICU, an expected average of 9 weeks. Note that registration and blood sampling only take place when a study drug is being administered
  level of ventilatory support, oxygen need (repetitive oxygenation index analyses), respiratory index and BPD development
EC50 of ibuprofen for patent ductus arteriosus (PDA) closure | Participants will be followed for the duration of admission to the NICU, an expected average of 9 weeks. Note that registration and blood sampling only take place when a study drug is being administered
  closure of PDA, significance of PDA

OTHER OUTCOMES:
Development of a minimally invasive Dried Blood Spot analysis method | Participants will be followed for the duration of admission to the NICU, an expected average of 9 weeks. Note that the validation of the Dried Blood Spot analysis can take place when a study drug is being administered
  The dried blood spot analyses will be validated to perform future pharmacokinetic studies in neonates. The measured concentration of the drugs in the dried blood spot samples will be compared with the concentration of the blood samples in the vial, which is the current validated standard method. The validity of the DBS method will be the endpoint.
Pharmacogenetic profile | Participants will be followed for the duration of admission to the NICU, an expected average of 9 weeks. Note that registration and blood sampling only take place when a study drug is being administered
  Influence of specific Single Nucleotide Polymorphisms on the genes that code for the enzymes that might be involved in the metabolism of the investigated drugs. Some of the related enzymes are CYP3A4 (sildenafil, midazolam, fentanyl), CYP2D6 (sildenafil), UGT (paracetamol), CYP2C9 and CYP2C19 (phenobarbital).

CONTACTS AND LOCATIONS:
Overall Officials: Ronald de Groot, MD, PhD, Study Director — Radboud University Medical Center; Dick Tibboel, MD, PhD, Study Chair — Erasmus Medical Center; David Burger, PharmD, PhD, Study Chair — Radboud University Medical Center
Locations (4):
- Netherlands (4):
  - MUMC, Maastricht
  - Radboud UMC, Nijmegen
  - Erasmus MC - Sophia Children's Hospital, Rotterdam
  - Maxima Medical Center, Veldhoven

REFERENCES:
- [Derived] Smit C, Engbers AGJ, Samiee-Zafarghandy S, van Donge T, Simons SHP, Flint RB, Pfister M, Knibbe CAJ, van den Anker JN. Oral Ibuprofen Is More Effective than Intravenous Ibuprofen for Closure of a Patent Ductus Arteriosus: Can Pharmacokinetic Modeling Help Us to Understand Why? Neonatology. 2023;120(1):81-89. doi: 10.1159/000526210. Epub 2022 Dec 9. PMID 36502794